CLINICAL TRIAL: NCT05257551
Title: Tempus Small Cell Lung Cancer Observational Study (Sculptor): A Tissue and Longitudinal Circulating Tumor DNA (ctDNA) Biomarker Profiling Study of Patients With Small Cell Lung Cancer (SCLC) Using Comprehensive Next-Generation Sequencing (NGS) Assays
Brief Title: Tempus Sculptor Study: Small Cell Lung Cancer (SCLC) Observational Study
Status: Recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-003
Record Dates: First submitted 2022-01-20; First posted 2022-02-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Cancer; Oncology; Observational; Genomic Profiling; Precision medicine; SCLC; Small Cell Lung Cancer; NGS; Biomarkers; ctDNA; Transcriptomics
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Small Cell Lung Cancer (SCLC): This protocol will include participants with newly diagnosed extensive stage (stage IV) small cell lung cancer with tissue collected from the primary lung tumor, or metastatic sites outside of the liver or biliary system.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention

SUMMARY:
The study is a non-interventional evaluation of participants with SCLC who will receive diagnostic and (where possible) post-progression tumor tissue profiling, alongside plasma ctDNA biomarker profiling in addition to their standard of care therapy and disease surveillance.

ELIGIBILITY:
The following are the inclusion criteria. Participants are eligible to be included in this study only if all the following criteria apply. The participant has/is:

* Histologically confirmed small cell lung cancer diagnosis
* Diagnosis made with excisional or core needle biopsy specimen (fine needle aspirate may be permitted with approval from the PI)
* Subjects must submit fresh or archived FFPE tumor sample to the central laboratory
* ECOG performance status of 0-2 at time of enrollment
* Planned extensive stage first-line therapy of etoposide plus carboplatin plus PD-L1 inhibitor (atezolizumab or durvalumab)
* Extensive stage disease at time of diagnosis
* Willing and able to provide informed consent
* Radiotherapy is permitted as long as there is measurable disease outside of the radiotherapy port

Participants will be excluded from the study if any of the following criteria apply. The participant has/is:

* History of prior systemic treatment of SCLC
* Prior diagnosis of non-small cell lung cancer is excluded if the cancer is diagnosed < 3 years prior to study entry. Additionally, the participant must be off all therapy for the NSCLC at the time of study entry.
* Mixed small cell and non-small cell histology
* Suspected metastatic cancer from other sites (i.e., those without a known or suspected lung primary diagnosis)
* Not willing to have additional blood samples collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This protocol targets patients with Small Cell Lung Cancer (SCLC)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
To determine if tumor tissue transcriptional subtypes can be detected | Up to 4 years
  To determine prospectively if SCLC tumor tissue transcriptional subtypes can be detected by Tempus|xT RNAseq
To characterize relationship between tissue transcriptional subtype and clinical outcomes | Up to 4 years
  To characterize the relationship between tissue transcriptional subtype and clinical outcomes for EP+PDL1-i therapy based on collection of longitudinal information from medical records

SECONDARY OUTCOMES:
To assess the potential for liquid biopsy in SCLC | Up to 4 years
  To use blood based assays to assess the complementarity of circulating biomarkers to tissue based methods
To test which tissue and sample variables confound gene expression subtypes | Up to 4 years
  To measure how variable transcriptional measurements are across tissue characteristics such as site of biopsy and type of biopsy

OTHER OUTCOMES:
To measure biomarkers of SCLC using the TEMPUS xT assay | Up to 4 years
  To measure specific biomarkers of SCLC subtypes and outcomes using the TEMPUS xT assay
To identify biomarkers and mechanisms of progression | Up to 4 years
  To identify biomarkers and mechanisms of progression from EP + PDL1-i therapy
To study progression free survival (PFS) and overall survival (OS) | Up to 4 years
  To study real-world PFS and OS as measured by the treating clinician

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Rhodes, MD, Principal Investigator — Tempus AI, Inc.
Locations (11):
- United States (11):
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - University of Colorado, Aurora, Colorado
  - Illinois Cancer Care, Peoria, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Englewood Health Medical Center, Englewood, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - TriHealth Cancer Institute, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Oklahoma Cancer Specialists and Research Institutes, Tulsa, Oklahoma
  - Cancer Care Association of York, York, Pennsylvania

REFERENCES:
- [Background] Ghosh S, Bilton JL. Torsion and infarction of the appendices epiploicae: Report of five cases. Dis Colon Rectum. 1968 Nov;11(6):457-61. doi: 10.1007/BF02616778. No abstract available. PMID 4972690
- [Background] Khondkarian OA, Zavalishin IA. [Several characteristics of "pyramid" insufficiency in lateral amyotrophic sclerosis]. Klin Med (Mosk). 1970 Sep;48(9):93-6. No abstract available. Russian. PMID 5497465
- [Background] van Beek EJ, Bakker AJ, Reekers JA. Pulmonary embolism: interobserver agreement in the interpretation of conventional angiographic and DSA images in patients with nondiagnostic lung scan results. Radiology. 1996 Mar;198(3):721-4. doi: 10.1148/radiology.198.3.8628860.
- [Background] Crowley E, Di Nicolantonio F, Loupakis F, Bardelli A. Liquid biopsy: monitoring cancer-genetics in the blood. Nat Rev Clin Oncol. 2013 Aug;10(8):472-84. doi: 10.1038/nrclinonc.2013.110. Epub 2013 Jul 9. PMID 23836314
- [Background] Drapkin BJ, Rudin CM. Advances in Small-Cell Lung Cancer (SCLC) Translational Research. Cold Spring Harb Perspect Med. 2021 Apr 1;11(4):a038240. doi: 10.1101/cshperspect.a038240. PMID 32513672
- [Background] Gay CM, Stewart CA, Park EM, Diao L, Groves SM, Heeke S, Nabet BY, Fujimoto J, Solis LM, Lu W, Xi Y, Cardnell RJ, Wang Q, Fabbri G, Cargill KR, Vokes NI, Ramkumar K, Zhang B, Della Corte CM, Robson P, Swisher SG, Roth JA, Glisson BS, Shames DS, Wistuba II, Wang J, Quaranta V, Minna J, Heymach JV, Byers LA. Patterns of transcription factor programs and immune pathway activation define four major subtypes of SCLC with distinct therapeutic vulnerabilities. Cancer Cell. 2021 Mar 8;39(3):346-360.e7. doi: 10.1016/j.ccell.2020.12.014. Epub 2021 Jan 21. PMID 33482121
- [Background] Goldman JW, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Garassino MC, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Thiyagarajah P, Jiang H, Paz-Ares L; CASPIAN investigators. Durvalumab, with or without tremelimumab, plus platinum-etoposide versus platinum-etoposide alone in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): updated results from a randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):51-65. doi: 10.1016/S1470-2045(20)30539-8. Epub 2020 Dec 4. PMID 33285097
- [Background] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Background] Kalemkerian GP, Loo BW, Akerley W, Attia A, Bassetti M, Boumber Y, Decker R, Dobelbower MC, Dowlati A, Downey RJ, Florsheim C, Ganti AKP, Grecula JC, Gubens MA, Hann CL, Hayman JA, Heist RS, Koczywas M, Merritt RE, Mohindra N, Molina J, Moran CA, Morgensztern D, Pokharel S, Portnoy DC, Rhodes D, Rusthoven C, Sands J, Santana-Davila R, Williams CC, Hoffmann KG, Hughes M. NCCN Guidelines Insights: Small Cell Lung Cancer, Version 2.2018. J Natl Compr Canc Netw. 2018 Oct;16(10):1171-1182. doi: 10.6004/jnccn.2018.0079. PMID 30323087
- [Background] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766
- [Background] Mahadevan NR, Knelson EH, Wolff JO, Vajdi A, Saigi M, Campisi M, Hong D, Thai TC, Piel B, Han S, Reinhold BB, Duke-Cohan JS, Poitras MJ, Taus LJ, Lizotte PH, Portell A, Quadros V, Santucci AD, Murayama T, Canadas I, Kitajima S, Akitsu A, Fridrikh M, Watanabe H, Reardon B, Gokhale PC, Paweletz CP, Awad MM, Van Allen EM, Lako A, Wang XT, Chen B, Hong F, Sholl LM, Tolstorukov MY, Pfaff K, Janne PA, Gjini E, Edwards R, Rodig S, Reinherz EL, Oser MG, Barbie DA. Intrinsic Immunogenicity of Small Cell Lung Carcinoma Revealed by Its Cellular Plasticity. Cancer Discov. 2021 Aug;11(8):1952-1969. doi: 10.1158/2159-8290.CD-20-0913. Epub 2021 Mar 11. PMID 33707236
- [Background] Ooki A, Maleki Z, Tsay JJ, Goparaju C, Brait M, Turaga N, Nam HS, Rom WN, Pass HI, Sidransky D, Guerrero-Preston R, Hoque MO. A Panel of Novel Detection and Prognostic Methylated DNA Markers in Primary Non-Small Cell Lung Cancer and Serum DNA. Clin Cancer Res. 2017 Nov 15;23(22):7141-7152. doi: 10.1158/1078-0432.CCR-17-1222. Epub 2017 Aug 29. PMID 28855354
- [Background] Rekhtman N. Lung neuroendocrine neoplasms: recent progress and persistent challenges. Mod Pathol. 2022 Jan;35(Suppl 1):36-50. doi: 10.1038/s41379-021-00943-2. Epub 2021 Oct 18. PMID 34663914
- [Background] Roper N, Velez MJ, Chiappori A, Kim YS, Wei JS, Sindiri S, Takahashi N, Mulford D, Kumar S, Ylaya K, Trindade C, Manukyan I, Brown AL, Trepel JB, Lee JM, Hewitt S, Khan J, Thomas A. Notch signaling and efficacy of PD-1/PD-L1 blockade in relapsed small cell lung cancer. Nat Commun. 2021 Jun 23;12(1):3880. doi: 10.1038/s41467-021-24164-y. PMID 34162872
- [Background] Rudin CM, Poirier JT, Byers LA, Dive C, Dowlati A, George J, Heymach JV, Johnson JE, Lehman JM, MacPherson D, Massion PP, Minna JD, Oliver TG, Quaranta V, Sage J, Thomas RK, Vakoc CR, Gazdar AF. Molecular subtypes of small cell lung cancer: a synthesis of human and mouse model data. Nat Rev Cancer. 2019 May;19(5):289-297. doi: 10.1038/s41568-019-0133-9. PMID 30926931
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Siravegna G, Marsoni S, Siena S, Bardelli A. Integrating liquid biopsies into the management of cancer. Nat Rev Clin Oncol. 2017 Sep;14(9):531-548. doi: 10.1038/nrclinonc.2017.14. Epub 2017 Mar 2. PMID 28252003
- [Background] Stewart CA, Gay CM, Xi Y, Sivajothi S, Sivakamasundari V, Fujimoto J, Bolisetty M, Hartsfield PM, Balasubramaniyan V, Chalishazar MD, Moran C, Kalhor N, Stewart J, Tran H, Swisher SG, Roth JA, Zhang J, de Groot J, Glisson B, Oliver TG, Heymach JV, Wistuba I, Robson P, Wang J, Byers LA. Single-cell analyses reveal increased intratumoral heterogeneity after the onset of therapy resistance in small-cell lung cancer. Nat Cancer. 2020 Apr;1:423-436. doi: 10.1038/s43018-019-0020-z. Epub 2020 Feb 17. PMID 33521652
- [Background] Tlemsani C, Pongor L, Elloumi F, Girard L, Huffman KE, Roper N, Varma S, Luna A, Rajapakse VN, Sebastian R, Kohn KW, Krushkal J, Aladjem MI, Teicher BA, Meltzer PS, Reinhold WC, Minna JD, Thomas A, Pommier Y. SCLC-CellMiner: A Resource for Small Cell Lung Cancer Cell Line Genomics and Pharmacology Based on Genomic Signatures. Cell Rep. 2020 Oct 20;33(3):108296. doi: 10.1016/j.celrep.2020.108296. PMID 33086069
- [Background] Zepp JA, Morrisey EE. Cellular crosstalk in the development and regeneration of the respiratory system. Nat Rev Mol Cell Biol. 2019 Sep;20(9):551-566. doi: 10.1038/s41580-019-0141-3. Epub 2019 Jun 19. PMID 31217577
- [Background] Zhang W, Girard L, Zhang YA, Haruki T, Papari-Zareei M, Stastny V, Ghayee HK, Pacak K, Oliver TG, Minna JD, Gazdar AF. Small cell lung cancer tumors and preclinical models display heterogeneity of neuroendocrine phenotypes. Transl Lung Cancer Res. 2018 Feb;7(1):32-49. doi: 10.21037/tlcr.2018.02.02. PMID 29535911
- [Background] Howlader, Nnam, A. M. Noone, Me Krapcho, D. Miller, A. Brest, M. Yu, J. Ruhl, et al. 2020."SEER Cancer Statistics Review, 1975--2017." National Cancer Institute.